CLINICAL TRIAL: NCT04363736
Title: A Phase-II, Open-Label, Randomized, Multicenter Study to Investigate the Pharmacodynamics, Pharmacokinetics, Safety, and Efficacy of 8 mg/kg or 4mg/kg Intravenous Tocilizumab in Patients With Moderate to Severe COVID-19 Pneumonia
Brief Title: A Study to Investigate Intravenous Tocilizumab in Participants With Moderate to Severe COVID-19 Pneumonia
Acronym: MARIPOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA42481
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TCZ 8 mg/kg (Active Comparator): Participants will receive intravenous (IV) tocilizumab (TCZ) at a dose of 8 mg/kg in addition to standard-of-care treatment.
  Interventions: Drug: Tociliuzumab
- TCZ 4 mg/kg (Experimental): Participants will receive IV tocilizumab (TCZ) at a dose of 4 mg/kg in addition to standard-of-care treatment.
  Interventions: Drug: Tociliuzumab

INTERVENTIONS:
Drug: Tociliuzumab — Participants will receive IV TCZ.

SUMMARY:
This study will assess the pharmacodynamics, pharmacokinetics, safety and efficacy of two different doses of tocilizumab (TCZ) in combination with standard-of-care (SOC) in hospitalized adult participants with moderate to severe COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria

* Hospitalization with COVID-19 pneumonia confirmed by a positive polymerase chain reaction (PCR) of any specimen [e.g., respiratory, blood, urine, stool, and other bodily fluids]) and evidence of pneumonia on chest X-ray or computed tomography scan
* For severe patients, SpO2 </= 93% or PaO2/FiO2 < 300 mmHg. If a participant is on supplemental oxygen with SpO2 > 93%, but desaturation </= to 93% on lower supplemental oxygen or ambient air is documented during screening, the inclusion criterion is met
* For moderate patients (those who do not qualify as severe based oxygen requirements), CRP > 2 x upper limit of normal (ULN) is required
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, as defined by the protocol
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined by the protocol

Exclusion Criteria

* Known severe allergic reactions to TCZ or other monoclonal antibodies
* Active tuberculosis (TB) infection
* Suspected active bacterial, fungal, viral, or other infection (besides SARS-CoV-2)
* Participants who are on a mechanical ventilator > 24 hours or extracorporeal membrane oxygenation (ECMO), in shock, or combination thereof with other organ failure requiring treatment in an ICU
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Receipt of oral anti-rejection or immunomodulatory drugs (including TCZ) within the past 3 months
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 10 x ULN detected within 24 hours at screening or at baseline (according to local laboratory reference ranges)
* Absolute neutrophil count (ANC) < 1000/uL at screening and baseline (according to local laboratory reference ranges)
* Platelet count < 50,000/uL at screening and baseline (according to local laboratory reference ranges)
* Pregnancy or breastfeeding, or positive pregnancy test at a predose examination
* Treatment with an investigational drug within 5 drug-elimination half-lives or 30 days (whichever is longer) of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- United States (24):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - St. Jude Medical Center, Fullerton, California
  - LAC + USC Medical Center, Los Angeles, California
  - USC Keck Medical Center of USC, Los Angeles, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - University of Maryland, Baltimore, Maryland
  - Renown Institute for Heart & Vascular Health, Reno, Nevada
  - St Joseph's Regional Medical Center, Wayne, New Jersey
  - SUNY Downstate Medical Center., Brooklyn, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny Health Network (Pittsburg PA), Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Kumar PN, Hernandez-Sanchez J, Nagel S, Feng Y, Cai F, Rabin J, Morse CG, Nadig NR, Ashraf O, Gotur DB, McComsey GA, Gafoor K, Perin P, Thornton SC, Stubbings W, Lin CJF, Tsai L. Safety and Efficacy of Tocilizumab 4 or 8 mg/kg in Hospitalized Patients With Moderate to Severe Coronavirus Disease 2019 Pneumonia: A Randomized Clinical Trial. Open Forum Infect Dis. 2021 Dec 4;9(1):ofab608. doi: 10.1093/ofid/ofab608. eCollection 2022 Jan. PMID 35024375
- [Derived] Tom J, Bao M, Tsai L, Qamra A, Summers D, Carrasco-Triguero M, McBride J, Rosenberger CM, Lin CJF, Stubbings W, Blyth KG, Carratala J, Francois B, Benfield T, Haslem D, Bonfanti P, van der Leest CH, Rohatgi N, Wiese L, Luyt CE, Kheradmand F, Rosas IO, Cai F. Prognostic and Predictive Biomarkers in Patients With Coronavirus Disease 2019 Treated With Tocilizumab in a Randomized Controlled Trial. Crit Care Med. 2022 Mar 1;50(3):398-409. doi: 10.1097/CCM.0000000000005229. PMID 34612846

RESULTS

PARTICIPANT FLOW:
Groups:
- TCZ 4 mg/kg: Participants received intravenous (IV) tocilizumab (TCZ) at a dose of 4 mg/kg in addition to standard-of-care treatment.
- TCZ 8 mg/kg: Participants received IV tocilizumab (TCZ) at a dose of 8 mg/kg in addition to standard-of-care treatment.
Period: Overall Study
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Started | 49 | 48
Completed | 30 | 35
Not Completed | 19 | 13
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 10 | 7
Not completed — Death | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (14.3) | 59.8 (14.6) | 58.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 27 | 30 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 15 | 26
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 20 | 13 | 33
  White | 15 | 23 | 38
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Day 0-28 (AUC0-d28) of Tocilizumab)
Time Frame: Days 0-28. Participants received a second dose within 8-24 hours after the initial infusion of TCZ at the discretion of the investigator upon clinically significant demonstration of worsening signs or symptoms.
Population: The PK population consisted of all randomized participants who received any amount of study drug with at least one valid pharmacokinetic (PK) result. Participants were analyzed according to treatment received.
Measure: Median (Full Range); unit: µg/mL*day
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 35 | 38
µg/mL*day
  One dose | 371 [196 to 1040] | 849 [471 to 1500]
  Two doses: number analyzed (Participants) | 12 | 9
  Two doses | 837 [592 to 1480] | 1330 [1130 to 1810]

2. Primary Outcome: Maximum Serum Concentration (Cmax) of Tocilizumab
Time Frame: Baseline - Day 60. Participants received a second dose within 8-24 hours after the initial infusion of TCZ at the discretion of the investigator upon clinically significant demonstration of worsening signs or symptoms.
Population: as for outcome 1
Measure: Median (Full Range); unit: µg/mL
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 35 | 38
µg/mL
  One dose | 82.2 [48.8 to 134] | 159 [101 to 234]
  Two doses: number analyzed (Participants) | 12 | 9
  Two doses | 150 [110 to 203] | 228 [198 to 363]

3. Primary Outcome: Clearance (CL) of Tocilizumab
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: L/day
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 35 | 38
L/day
  One dose | 0.451 [0.261 to 0.697] | 0.487 [0.179 to 1.16]
  Two doses: number analyzed (Participants) | 12 | 9
  Two doses | 0.468 [0.327 to 0.701] | 0.629 [0.376 to 1.02]

4. Primary Outcome: Volume of the Central Compartment (Vc) of Tocilizumab
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: L
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 35 | 38
L
  One dose | 4.14 [2.47 to 7.11] | 4.34 [3.08 to 7.88]
  Two doses: number analyzed (Participants) | 12 | 9
  Two doses | 4.2 [2.54 to 5.17] | 4.57 [3.59 to 7.27]

5. Primary Outcome: Serum Concentration of C-reactive Protein (CRP) Following Administration of IV TCZ
Time Frame: Baseline - Day 60
Population: Modified intent-to-treat population (mITT): All randomized participants who received any amount of study drug. Participants are analyzed according to the treatment assigned at randomization.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
mg/L
  Baseline: number analyzed (Participants) | 45 | 42
  Baseline | 125.04 (121.5) | 115.77 (128.7)
  Day 1 - 15 min post-dose: number analyzed (Participants) | 43 | 37
  Day 1 - 15 min post-dose | 124.67 (118.8) | 109.19 (134.4)
  Day 1 - pre-dose 2nd infusion: number analyzed (Participants) | 10 | 6
  Day 1 - pre-dose 2nd infusion | 123.49 (68.0) | 118.83 (45.1)
  Day 1 - 15 min post-dose 2nd infusion: number analyzed (Participants) | 12 | 6
  Day 1 - 15 min post-dose 2nd infusion | 116.89 (62.4) | 112.97 (53.4)
  Day 2 - 24 hours post-dose: number analyzed (Participants) | 41 | 38
  Day 2 - 24 hours post-dose | 85.75 (133.1) | 86.01 (124.2)
  Day 3: number analyzed (Participants) | 40 | 37
  Day 3 | 41.56 (129.6) | 39.17 (134.8)
  Day 7: number analyzed (Participants) | 33 | 30
  Day 7 | 7.27 (145.1) | 5.62 (188.3)
  Day 14: number analyzed (Participants) | 19 | 21
  Day 14 | 4.42 (554.8) | 0.87 (95.0)
  Day 21: number analyzed (Participants) | 10 | 17
  Day 21 | 3.73 (552.5) | 1.75 (1681.6)
  Day 28: number analyzed (Participants) | 9 | 19
  Day 28 | 3.01 (483.0) | 2.57 (2251.1)
  Day 35: number analyzed (Participants) | 4 | 8
  Day 35 | 2.12 (234.5) | 11.25 (1543.9)
  Day 60: number analyzed (Participants) | 13 | 19
  Day 60 | 2.41 (256.0) | 1.61 (154.1)

6. Primary Outcome: Serum Concentration of Ferritin Following Administration of IV TCZ
Time Frame: Baseline - Day 60
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
pmol/L
  Baseline: number analyzed (Participants) | 42 | 38
  Baseline | 2081.46 (162.4) | 1821.19 (174.0)
  Day 2 - 24 hours post-dose: number analyzed (Participants) | 19 | 20
  Day 2 - 24 hours post-dose | 2282.62 (191.3) | 1938.19 (154.6)
  Day 3: number analyzed (Participants) | 37 | 34
  Day 3 | 2016.10 (128.0) | 2060.41 (131.2)
  Day 7: number analyzed (Participants) | 24 | 29
  Day 7 | 1760.82 (170.3) | 1494.76 (86.7)
  Day 14: number analyzed (Participants) | 16 | 20
  Day 14 | 1108.34 (127.2) | 720.66 (102.3)
  Day 21: number analyzed (Participants) | 11 | 16
  Day 21 | 754.24 (138.4) | 558.57 (119.0)
  Day 28: number analyzed (Participants) | 9 | 18
  Day 28 | 393.46 (139.3) | 519.51 (139.0)
  Day 35: number analyzed (Participants) | 4 | 8
  Day 35 | 309.23 (105.5) | 291.24 (66.5)
  Day 60: number analyzed (Participants) | 13 | 17
  Day 60 | 282.85 (148.7) | 246.17 (171.4)

7. Primary Outcome: Serum Concentration of Soluble Interleukin-6 Receptor (sIL-6R) Following Administration of IV TCZ
Time Frame: Baseline - Day 60
Population: Modified intent-to-treat population (mITT): All randomized participants who received any amount of study drug. Participants are analyzed according to the treatment assigned at randomization. Participants at Day 2 15-min post-dose were those that received a second dose of TCZ and had PK taken after that second dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/L
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
ng/L
  Baseline: number analyzed (Participants) | 45 | 43
  Baseline | 35869.87 (29.1) | 35331.04 (31.3)
  Day 1 - 15 min post-dose: number analyzed (Participants) | 46 | 44
  Day 1 - 15 min post-dose | 47037.59 (56.1) | 40928.43 (46.4)
  Day 2 - 15 min post-dose: number analyzed (Participants) | 2 | 1
  Day 2 - 15 min post-dose | 80880.16 (24.9) | 44300.00 (NA) — CV not available for a single value.
  Day 2 - 24 hours post-dose: number analyzed (Participants) | 40 | 38
  Day 2 - 24 hours post-dose | 97280.14 (31.3) | 90057.53 (28.8)
  Day 3: number analyzed (Participants) | 40 | 38
  Day 3 | 139128.70 (26.5) | 139528.82 (30.3)
  Day 7: number analyzed (Participants) | 33 | 31
  Day 7 | 261637.28 (30.2) | 263899.86 (26.7)
  Day 14: number analyzed (Participants) | 19 | 22
  Day 14 | 258484.08 (52.3) | 339661.18 (19.6)
  Day 21: number analyzed (Participants) | 11 | 18
  Day 21 | 162025.68 (73.1) | 265981.84 (49.1)
  Day 28: number analyzed (Participants) | 9 | 20
  Day 28 | 82508.76 (102.6) | 162795.31 (106.0)
  Day 35: number analyzed (Participants) | 5 | 9
  Day 35 | 80425.91 (138.7) | 144868.00 (105.4)
  Day 60: number analyzed (Participants) | 15 | 18
  Day 60 | 36049.91 (21.7) | 34258.34 (22.2)

8. Primary Outcome: Serum Concentration of Interleukin-6 (IL-6) Following Administration of IV TCZ
Time Frame: Baseline - Day 60
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/L
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
ng/L
  Day 1 - 15 min post-dose: number analyzed (Participants) | 46 | 44
  Day 1 - 15 min post-dose | 336.99 (248.8) | 325.96 (236.4)
  Day 2 - 15 min post-dose: number analyzed (Participants) | 2 | 1
  Day 2 - 15 min post-dose | 292.69 (159.8) | 638.00 (NA) — CV not available for a single value.
  Day 2 - 24 hours post-dose: number analyzed (Participants) | 41 | 38
  Day 2 - 24 hours post-dose | 733.99 (226.5) | 757.17 (172.4)
  Day 3: number analyzed (Participants) | 40 | 37
  Day 3 | 748.82 (394.2) | 743.84 (263.0)
  Day 7: number analyzed (Participants) | 30 | 31
  Day 7 | 545.44 (315.9) | 589.21 (429.0)
  Day 14: number analyzed (Participants) | 18 | 22
  Day 14 | 234.88 (332.2) | 125.64 (345.9)
  Day 21: number analyzed (Participants) | 11 | 17
  Day 21 | 49.16 (482.7) | 91.86 (465.9)
  Day 28: number analyzed (Participants) | 9 | 19
  Day 28 | 5.73 (NA) — Geometric CV not reported when more than 1/3 of post-dose PK samples are below the limit of quantitation. | 28.66 (371.7)
  Day 35: number analyzed (Participants) | 5 | 8
  Day 35 | 7.68 (361.9) | 39.79 (503.0)
  Day 60: number analyzed (Participants) | 15 | 17
  Day 60 | 2.52 (NA) — Geometric CV not reported when more than 1/3 of post-dose PK samples are below the limit of quantitation. | 2.28 (NA) — Geometric CV not reported when more than 1/3 of post-dose PK samples are below the limit of quantitation.

9. Secondary Outcome: Pecentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to Day 60
Population: The safety population included all randomized participants who received any amount of study drug, with participants analyzed according to the treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
Percentage of Participants | 57.1 | 45.8

10. Secondary Outcome: Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-CoV-2) (COVID-19) Viral Load Over Time
Time Frame: Baseline - Day 60
Population: as for outcome 9
Measure: Median (Full Range); unit: copies/µL
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
copies/µL
  Baseline: number analyzed (Participants) | 46 | 46
  Baseline | 30.56 [0.1 to 14458.9] | 8.51 [0.1 to 132429.0]
  Day 2: number analyzed (Participants) | 45 | 41
  Day 2 | 8.38 [0.1 to 6328.1] | 7.90 [0.1 to 264252.7]
  Day 3: number analyzed (Participants) | 40 | 40
  Day 3 | 3.82 [0.1 to 338006.1] | 4.46 [0.1 to 135875.7]
  Day 4: number analyzed (Participants) | 35 | 32
  Day 4 | 2.44 [0.1 to 17142.1] | 2.73 [0.1 to 159013.2]
  Day 5: number analyzed (Participants) | 31 | 26
  Day 5 | 8.74 [0.1 to 2930.4] | 5.39 [0.1 to 59216.3]
  Day 6: number analyzed (Participants) | 24 | 23
  Day 6 | 0.91 [0.1 to 41683.2] | 2.56 [0.1 to 13318.7]
  Day 7: number analyzed (Participants) | 29 | 28
  Day 7 | 0.49 [0.1 to 11609.3] | 1.47 [0.1 to 14185.5]
  Day 10: number analyzed (Participants) | 19 | 16
  Day 10 | 2.56 [0.1 to 149.3] | 0.59 [0.1 to 556.2]
  Day 14: number analyzed (Participants) | 18 | 23
  Day 14 | 0.14 [0.1 to 26.5] | 0.18 [0.1 to 436.5]
  Day 21: number analyzed (Participants) | 13 | 18
  Day 21 | 0.1 [0.1 to 39.6] | 0.12 [0.1 to 56.4]
  Day 28: number analyzed (Participants) | 10 | 21
  Day 28 | 0.16 [0.1 to 3.6] | 0.12 [0.1 to 3.4]
  Day 35: number analyzed (Participants) | 4 | 5
  Day 35 | 0.1 [0.1 to 0.2] | 0.12 [0.1 to 5.6]
  Day 45: number analyzed (Participants) | 2 | 4
  Day 45 | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  Early withdrawal: number analyzed (Participants) | 0 | 1
  Early withdrawal |  | 0.1 [0.1 to 0.1]
  Day 60: number analyzed (Participants) | 10 | 17
  Day 60 | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.3]

11. Secondary Outcome: Time to Real-Time Polymerase Chain Reaction (RT-PCR) Virus Negativity
Description: Time to Real-Time Polymerase Chain Reaction (RT-PCR) virus negativity was defined as the number of days from the first dose of study drug to when a negative RT-PCR SARS-CoV-2 assessment result was observed. Results are presented as a cumulative incidence function (CIF) with death as a competing risk.
Time Frame: Up to Day 28
Population: Only participants with at least one virology assessment were included in the analysis.
Measure: Number; unit: Probability
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
Probability
  CIF for event on Day 7: number analyzed (Participants) | 48 | 48
  CIF for event on Day 7 | 0.3389 | 0.2874
  CIF for death on Day 7: number analyzed (Participants) | 48 | 48
  CIF for death on Day 7 | 0.0665 | 0.0000
  CIF for event on Day 14: number analyzed (Participants) | 48 | 48
  CIF for event on Day 14 | 0.5068 | 0.5727
  CIF for death on Day 14: number analyzed (Participants) | 48 | 48
  CIF for death on Day 14 | 0.1024 | 0.0884
  CIF for event on Day 21: number analyzed (Participants) | 48 | 48
  CIF for event on Day 21 | 0.5068 | 0.5727
  CIF for death on Day 21: number analyzed (Participants) | 48 | 48
  CIF for death on Day 21 | 0.1497 | 0.1280
  CIF for event on Day 28: number analyzed (Participants) | 48 | 48
  CIF for event on Day 28 | 0.5730 | 0.6327
  CIF for death on Day 28: number analyzed (Participants) | 48 | 48
  CIF for death on Day 28 | 0.3420 | 0.1793

12. Secondary Outcome: Proportion of Participants With Any Post-Treatment Infection
Time Frame: Up to Day 60
Measure: Number; unit: Percentage of Participants
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
Number analyzed (Participants) | 49 | 48
Percentage of Participants
  COVID-19 pneumonia | 6.1 | 2.1
  Sepsis | 2.0 | 4.2
  Septic shock | 2.0 | 4.2
  Pneumonia | 2.0 | 2.1
  Urinary tract infection | 2.0 | 2.1
  Abscess limb | 2.0 | 0
  Atypical pneumonia | 2.0 | 0
  Pneumonia bacterial | 2.0 | 0
  Pneumonia klebsiella | 2.0 | 0
  Pneumonia streptococcal | 2.0 | 0
  Staphylococcal infection | 2.0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 60
Arm/Group | TCZ 4 mg/kg | TCZ 8 mg/kg
All-Cause Mortality (participants affected / at risk) | 8/49 | 6/48
Serious Adverse Events (participants affected / at risk) | 15/49 | 12/48
Other Adverse Events (participants affected / at risk) | 4/49 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCZ 4 mg/kg (N=49) | TCZ 8 mg/kg (N=48)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Sputum culture positive (Investigations) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 4 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCZ 4 mg/kg (N=49) | TCZ 8 mg/kg (N=48)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT04363736/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04363736/SAP_001.pdf